CLINICAL TRIAL: NCT03961685
Title: The CALM Study: Cancer Activity and Lifestyle Measurement Study
Brief Title: Cancer Activity and Lifestyle Measurement Study
Acronym: CALM
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Carol S. Kennedy Professor, Ohio State University
Other Study IDs: 2017C0165
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The CALM Study is an observational study to investigate the associations of linoleic acid levels in the blood, diet, activity, and lifestyle factors with measures of muscle strength, muscle function and overall outcomes for postmenopausal breast cancer patients treated with anthracycline chemotherapy.

DETAILED DESCRIPTION:
The CALM Study is a prospective study to determine the effects of adjuvant chemotherapy on cardiolipin profiles in relationship to cardiac and skeletal muscle function in breast cancer patients before and after 1 cycle of anthracycline therapy. Patients will undergo blood sampling and imaging of the heart and skeletal muscle at two Clinical Visits. The two visits, Baseline and study completion (Post-1 cycle anthracycline) will occur approximately ~4 weeks apart.

The driving hypothesis is that anthracycline reduces linoleic acid-rich cardiolipin with associated decline of cardiac and skeletal muscle measures. By coupling cardiac and skeletal muscle changes with cardiolipin markers reflective of dietary linoleic acid, this work will advance inexpensive and highly accessible therapies to preserve functional capacity and diminish adverse outcomes in cancer patients. Breast cancer patients (stages I-III) receiving anthracycline will be prospectively evaluated to achieve the following aims:

Aim 1: Measure the baseline relationships between cardiolipin status and magnetic resonance-based measures of cardiac and skeletal muscle physiology in breast cancer patients. Hypothesis 1a: Higher cardiolipin is related to better cardiac structure and function. Hypothesis 1b: Higher cardiolipin is associated with higher skeletal muscle mass and mitochondrial capacity in women with breast cancer prior to starting anthracycline therapy. Hypothesis 1c: Dietary linoleic acid modifies the relationships between cardiolipin and cardiac or skeletal muscle measures.

Aim 2: Assess chemotherapy-induced changes in cardiolipin composition, cardiac and skeletal muscle physiology. Hypothesis 2a: Change in skeletal muscle function and cardiac function together better predict worse functional capacity after completion of a course of anthracycline therapy for breast cancer compared to change of either skeletal or cardiac function alone. Hypothesis 2b: Cardiolipin levels decrease significantly from baseline in women who have completed one cycle of anthracycline therapy for breast cancer. Hypothesis 2c: Dietary linoleic acid modifies the effects of anthracycline on cardiolipin and cardiac or skeletal muscle physiology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-II breast cancer, adjuvant or neoadjuvant anthracycline therapy

Exclusion Criteria:

* current smoker, under medical supervision for any other type of cancer, prior history of malignancies, infection requiring antibiotics in the last 3 months, diagnosis of hear disease or previous heart attach, stroke, or heart surgery, pacemaker or defibrillator, cardiac edema, autoimmune or inflammatory disease, current use of hormone replacement therapy, liver diseases, kidney diseases or failure, digestive diseases, pulmonary diseases or edema, diabetes, severe claustrophobia and/or metal implants preventing MRI measurement, orthopedic diagnoses prevent mobility, mitochondrial diseases, any other condition that would impede or be contraindicated for study assessments

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women ≥25 and < 70 years with stage I-III breast cancer who have adjuvant or neoadjuvant planned AC treatment will be screened for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiac Magnetic Resonance from baseline to study completion, an average of 3 weeks) | Baseline and study completion, an average of 3 weeks
  Measurement of Cardiac Functions using Magnetic Resonance Imaging (MRI)
Change in Skeletal Muscle 31Phosphorous Magnetic Resonance Spectroscopy (P-MRS) from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measurement of energy recovery and fat content of the calf muscle
Change in Peripheral Blood Mononuclear Cell Cardiolipin from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measurement of a phospholipid in the mitochondrial membrane of white blood cells

SECONDARY OUTCOMES:
Change in Habitual and recent dietary intake from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measurement of dietary intake in the past month using Dietary History Questionnaire and recent intake will be measured using 24-hour recall
Change in Physical Activity Questionnaires from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  two questionnaire will be used to measure physical activity and leisure time activity
Change in Breast Cancer Prevention Trial (BCPT) symptoms from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  BCPT symptoms questionnaire measures symptoms related to breast cancer treatment
Change in Fatigue Questionnaire from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measures fatigue in breast cancer patients
Change in Short form Health Survey (SF-36) Questionnaire from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measures general physical functioning and well-being
Change in Sleep Disturbance Questionnaire from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Assesses sleep quality and sleep-related impairments
Change in Linoleic Acid in the blood from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Linoleic acid levels in the plasma and erythrocytes
Change in Dual-Energy X-Ray Absorptiometry (DEXA) from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measures body composition (adipose and muscle mass)
Change in MRI liver lipid content from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measurement of Liver Lipid content using Magnetic Resonance Imaging (MRI)

OTHER OUTCOMES:
Change in Body Mass Index (BMI) from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Indirect measure of body composition using weight and height
Change in Omega-3 Intake Checklist from baseline to study completion, an average of 3 weeks | Baseline and study completion, an average of 3 weeks
  Measure the amount of omega-3 fatty acid consumed in the diet

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Clinical Research Center (Davis Medical Research Center), Columbus, Ohio, United States

REFERENCES:
- [Derived] Marris KE, Cole RM, Addison D, Ruz P, Sparagna G, Ni A, Belury MA. The Relationship Between Blood Lipidomics and Cardiotoxic Injury Following Acute Exposure to Anthracycline Chemotherapy in Women With Breast Cancer: A Feasibility Study. Curr Dev Nutr. 2025 Sep 4;9(10):107552. doi: 10.1016/j.cdnut.2025.107552. eCollection 2025 Oct. PMID 41069420